CLINICAL TRIAL: NCT07036588
Title: Modified Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial(PALARC 02)
Brief Title: PARLAR-02 Trial：Modified Transanal Drainage Tube Use for Preventing Anastomotic Leakage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Department head, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TDT20250616
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mTDT Group (Experimental): Patients will undergo elective laparoscopic/robotic low anterior resection and will be subjected to a modified perianal drainage tube intervention.
  Interventions: Device: Modified Transanal Drainage Tube
- Non-mTDT Group (No Intervention): Patients will undergo elective laparoscopic/robotic low anterior resection and will NOT be subjected to a modified perianal drainage tube intervention.

INTERVENTIONS:
Device: Modified Transanal Drainage Tube — Patients with rectal adenocarcinoma will undergo elective laparoscopic/robotic low anterior resection. After the anastomosis is completed and the air leak test is confirmed to be negative, a modified TDT (occlusive balloon catheter) will be inserted. The balloon will be placed 5 cm above the anastomosis and filled under laparoscopic visualization (approximately 25 ml) to slightly dilate the intestinal lumen and occlude the intestinal cavity (under laparoscopic monitoring to ensure it does not affect the blood supply of the intestine). The external part of the tube will be sutured to the perianal skin and further secured with a 3M transparent dressing on the outside. It will be connected to a drainage bag (with an inner diameter greater than 8 mm) and left in place for 7 days, or until the drainage function is lost due to obvious defecation around the anal tube, at which point the catheter will be removed.
  Arms: mTDT Group

SUMMARY:
Surgical resection remains the primary treatment for rectal cancer, but the postoperative incidence of anastomotic leakage (AL) is relatively high. AL not only increases the medical burden on patients, prolongs hospital stays, raises the need for secondary surgery, and elevates perioperative mortality, but also increases the long-term risk of local recurrence and reduces survival rates. There is an urgent need for a simple, effective treatment method that minimizes the burden on patients to prevent anastomotic leakage.

The preoperative placement of a transanal drainage tube (TDT) is believed to effectively drain gas and feces from the intestinal lumen, thereby reducing intestinal pressure and alleviating tension at the anastomotic site, thus preventing AL. Previous studies have shown that traditional drainage tubes cannot effectively prevent leakage. Given the limitations of existing research on traditional TDTs, we plan to use a modified TDT (which allows postoperative irrigation and utilizes a balloon to block feces from adversely affecting the anastomosis) to conduct a randomized, parallel-controlled trial. This study aims to further investigate the role of the modified TDT in preventing and treating anastomotic leakage following rectal surgery

DETAILED DESCRIPTION:
Patients were randomly assigned to two groups: the modified-TDT group and the non-modified-TDT group. Randomization was achieved using a computer-generated random number sequence allocation. To ensure all intraoperative decisions made by the surgeon remained unaffected by group assignment, surgeon allocation concealment was implemented : Surgeons were only informed of the group assignment and implemented the intervention according to the randomization result after completing the intestinal anastomosis and deciding whether to create a diverting stoma (DS) during the surgery. All surgical procedures strictly adhered to the guidelines for the diagnosis and treatment of colorectal cancer and the principles of total mesorectal excision (TME). Preservation of the left colic artery (LCA) was determined by the surgeon based on their experience and assessment of the patient's condition. Upon completion of the anastomosis, the surgeon decided on DS construction based on an assessment of risk factors for anastomotic leakage (AL). Pelvic drainage was utilized in all cases in this study.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma (confirmed by pathology);
* Tumor location: The lower edge is ≤10 cm from the anal verge;
* Age: ≥18 and ≤80 years old;
* ASA ≤3 ;
* After assessment, laparoscopic/robotic sphincter - preserving surgery for rectal cancer is feasible;
* T2 - 4N0 - 3M0~T0 - 1N1 - 3M0 & non- local recurrence;
* Signed informed consent form;
* Able to understand the risks of participating in the trial.

Exclusion Criteria:

* Emergency surgery;
* Presence of multiple primary colorectal cancers;
* History of long - term use of immunosuppressants or corticosteroids;
* Patients with severe mental illness or uncontrolled infection before surgery;
* Pregnant or breastfeeding women;
* Bowel obstruction before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AL | The time frame is from the completion of the surgery to the 30th day after the surgery.
  The incidence of total anastomotic leakage within 30 days after surgery

SECONDARY OUTCOMES:
Grades of AL | The time frame is from the completion of the surgery to the 30th day after the surgery.
  Classification of anastomotic leakage: Grade A is asymptomatic and detected by imaging only; Grade B requires specific interventions but not surgical treatment; Grade C requires surgical treatment.
Incidence of anastomosis-related complications | The time frame is from patient discharge to the 12th month after surgery.
  The overall incidence of anastomosis-related complications within 12 months after surgery.
3y-DFS AND LRR | The time frame is from patient discharge to the third year after surgery.
  Three-year disease-free survival (DFS) and local recurrence rate.
Perianal pain assessment score | Measurement Time Points: Postoperative Day 1, Day 3, and Day 5
  Numerical Rating Scale (NRS) [0-10 scale]: No pain (0); Mild pain (1-3); Moderate pain (4-6); Severe pain (7-10)

CONTACTS AND LOCATIONS:
Overall Officials: WeiDong Tong, Principal Investigator — Army Medical University, China
Locations (1):
- Army Medical Center (Daping Hospital), Yuzhong, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao S, Zhang L, Gao F, Wu M, Zheng J, Bai L, Li F, Liu B, Pan Z, Liu J, Du K, Zhou X, Li C, Zhang A, Pu Z, Li Y, Feng B, Tong W. Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Laparoscopic Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1151-1158. doi: 10.1001/jamasurg.2021.4568. PMID 34613330